CLINICAL TRIAL: NCT06290687
Title: Phase II Trial on the Safety and Efficacy of Partial Cystectomy and Extended Pelvic Lymph Node Dissection With Standard of Care Perioperative Systemic Therapy in the Management of Muscle-Invasive Bladder Cancer (PRESERVE Trial)
Brief Title: Partial Cystectomy & Extended Pelvic Lymph Node Dissection With SOC Perioperative Systemic Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASE5824
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Malignant Neoplasm of Bladder; Muscle Invasive Bladder Carcinoma
Keywords: Partial cystectomy; Pelvic Lymph Node Dissection
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Neoadjuvant Therapy; Cystectomy

STUDY DESIGN:
Intervention Model Description: This is a single-center, prospective, phase II trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cisplatin Eligible Participants (Experimental): Participants who are deemed eligible for cisplatin-based NAC will undergo:
  * Standard of care neoadjuvant systemic therapy (currently cisplatin-based chemotherapy in cisplatin-eligible participants)
  * Partial cystectomy with extended pelvic lymph node dissection
  * Standard of care adjuvant systemic therapy in eligible patients
  Interventions: Drug: Neoadjuvant Chemotherapy; Procedure: Partial cystectomy with Extended pelvic lymph node dissection; Drug: Adjuvant systemic therapy
- Cisplatin Ineligible Participants (Experimental): Participants who are deemed ineligible for cisplatin-based NAC will undergo:
  * Partial cystectomy with extended pelvic lymph node dissection
  * Standard of care adjuvant systemic therapy in eligible participants
  Interventions: Procedure: Partial cystectomy with Extended pelvic lymph node dissection; Drug: Adjuvant systemic therapy

INTERVENTIONS:
Drug: Neoadjuvant Chemotherapy — Standard of care neoadjuvant systemic therapy is currently cisplatin-based chemotherapy in cisplatin-eligible participants. Participants will start treatment within 60 days of Transurethral Resection of Bladder Tumor. Regimens may include:
  * Cisplatin - Gemcitabine (Gem/Cis)
  * Dose Dense Methotrexate - Vinblastine - Adriamycin - Cisplatin (MVAC)
  Arms: Cisplatin Eligible Participants
Procedure: Partial cystectomy with Extended pelvic lymph node dissection — Partial cystectomy will then be performed using the surgical technique at the discretion of the treating Urologic Oncologist. Extended pelvic lymphadenectomy will then be performed at the discretion of the treating Urologic Oncologist. Surgery will be performed within 60 days of Transurethral Resection of Bladder Tumor for Cisplatin-ineligible participants. Surgery will be performed within 60 days of completing neoadjuvant chemotherapy for Cisplatin-eligible participants.
Drug: Adjuvant systemic therapy — Standard of care adjuvant systemic therapy in eligible participants. The choice of adjuvant systemic therapy will be left to the discretion of the treating Medical Oncologist but must fall within the SOC as outlined in NCCN guidelines.

SUMMARY:
The goal of this clinical trial is to determine if a partial cystectomy with extended pelvic lymph node removal will be effective at treating Muscle-Invasive Bladder Cancer instead of a complete cystectomy with extended pelvic lymph node removal. This clinical trial aims to determine the safety and oncologic efficacy of the intervention, and to examine patient-reported quality of life outcomes in participants. Participants will receive the standard pre-surgery treatment for approximately 4 to 6 weeks. After the pre-surgery treatment is completed, participants will undergo a partial cystectomy with extended pelvic lymph node dissection. After surgery, participants will receive adjuvant systemic therapy.

DETAILED DESCRIPTION:
Radical cystectomy (surgical removal of the bladder) with pelvic lymph node dissection and urinary diversion, with neoadjuvant chemotherapy in eligible participants, is the standard of care in participants with muscle-invasive bladder cancer (MIBC). While this has demonstrated efficacy in the treatment of MIBC, it has risk of perioperative morbidity and impacts quality of life. Partial cystectomy (surgical removal of a portion of the bladder) is one option for bladder-sparing treatment of select bladder cancer participants and is included in the National Comprehensive Cancer Network bladder cancer treatment guidelines. This treatment has the advantage of less invasive treatment with a lower risk of surgical complication and better health-related quality of life (HRQOL) while providing pathologic staging, however there are limited data on outcomes with this treatment, especially patient-reported HRQOL outcomes. Additionally, much of the existing literature on efficacy of this treatment predates the use of advanced imaging in preoperative staging and advances in surgical technique including use of minimally-invasive surgical approaches and enhanced-recovery post-operative care paths. Given these limitations in the existing literature, the aim of this clinical trial is to examine the safety and efficacy and HRQOL outcomes of partial cystectomy with extended pelvic lymph node dissection, with standard of care perioperative systemic therapy in eligible participants.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically confirmed urothelial carcinoma of the bladder, clinical stage T2-3N0M0. Micropapillary, glandular, squamous, and sarcomatoid histologic variants of urothelial carcinoma are allowed.
* Subjects must have unifocal or limited multifocal disease amenable to complete surgical resection with partial cystectomy, as judged by the treating urologic oncologist.
* Age >18 years. Because of the rarity of this disease and limited data on treatment efficacy in subjects 18 years of age, children are excluded from this study.
* Performance status - Karnofsky Performance Status ≥70 or Eastern Cooperative Oncology Group (ECOG) performance status Grade 0 or 1.
* Subjects must have normal organ and marrow function as defined below:

  * Total bilirubin within normal limits
  * AST (SGOT) ≤ 2.5 X institutional upper limit of normal
  * ALT (SGPT) ≤ 2.5 X institutional upper limit of normal
  * Bone marrow:

    * Absolute neutrophil count (ANC) ≥ 1,500/mm3
    * Platelet count ≥ 80,000/mm3, Hemoglobin ≥ 9.0 g/dL
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.
* Subjects must have tumor less than or equal to 5 cm in largest dimension as assessed radiographically.
* Treatment naive for MIBC.

Exclusion Criteria:

* Presence of hydronephrosis.
* Presence of multifocal disease that is not amenable to complete resection with partial cystectomy.
* Presence of distant carcinoma in situ.
* Presence of clinical N+ or M+ disease.
* Presence of cT4+ disease.
* Non-urothelial histology.
* Concurrent upper tract (ureter or renal pelvis) or urethral urothelial carcinoma.
* Subjects who are not surgical candidates due to competing medical comorbidities or who refuse surgical treatment.
* Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (eg, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2026-01-29 (Estimated); Study Completion 2027-01-29 (Estimated)

PRIMARY OUTCOMES:
Recurrence-Free Survival (RFS) | Up to 24 months from date of post-surgery baseline scan
  Recurrence-Free Survival (RFS) is defined as the time from post-surgery baseline scan (revealing no recurrent/metastatic disease) until the first occurrence of either local or distant recurrence as assessed by CT or MRI and/or biopsy. The primary outcome of distant RFS will be assessed via Kaplan-Meier analysis

SECONDARY OUTCOMES:
Presence of Post-operative Complications | At 90 days after surgery
  The Clavien-Dindo classification will measure post-operative complications. The Clavien-Dindo Classification of Post-operative Complications is a tool to assess complications following surgical treatment. This tool ranks complications on a scale of seven levels, with level 1 being the least complicated and 7 being the worst complication resulting in death. The average classification at 90 days will be assessed and reported.
Median Bladder RFS | Up to 24 months from date of post-surgery baseline scan
  The median duration of bladder recurrence-free survival at 2 years.
Median Muscle-Invasive Bladder RFS | Up to 24 months from date of post-surgery baseline scan
  The median duration of muscle-invasive bladder recurrence-free survival at 2 years.
Median Bladder-Intact Survival | Up to 24 months from date of post-surgery baseline scan
  The median duration of bladder-intact survival at 2 years.
Median Cancer-Specific Survival | Up to 24 months from date of post-surgery baseline scan
  The median duration of cancer-specific survival at 2 years.
Changes in Genitourinary-specific HRQoL | Up to 24 months from date of post-surgery baseline scan
  The mean changes in Genitourinary-specific HRQoL will be reported. The HRQoL survey is composed of five functional scales (physical, role, emotional, cognitive, and social functioning), three symptom scales (fatigue, nausea and vomiting, pain), a global health status/QoL, and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The scales and single-item measures range from 0 - 100, with higher values representing a higher response level.

CONTACTS AND LOCATIONS:
Overall Officials: Nima Almassi, MD, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center
Locations (1):
- Glickman Urological and Kidney Institute, Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No